CLINICAL TRIAL: NCT01899365
Title: An Incitative Multifaceted PROcedure for Pneumococcal Vaccination at the Emergency Department; A Multicenter Prospective Randomized Open Trial The IMPROVED Project
Brief Title: An Incitative Multifaceted PROcedure for Pneumococcal Vaccination at the Emergency Department
Acronym: IMPROVED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Collaborators: Centre Scientifique de Monaco (Other); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-09; 2013-A00943-42 (Other: ANSM)
Record Dates: First submitted 2013-07-04; First posted 2013-07-15 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2017-10

CONDITIONS: Pneumococcal Infections
Keywords: anti-pneumococcal vaccination; information; emergency department
MeSH Terms: conditions — Pneumococcal Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Multifaceted: * brief structured interview with the physician about pneumococcal risk and vaccination,
  * information sheet delivered to patients with explanation about risk and benefit of APV,
  * letter given to patient for his/her general practitioner stating that the patient is at-risk for pneumococcal infection and could benefit of APV,
  * 3 SMS every 2 weeks to remind patients talking of pneumococcal risk with general practitioner.
- Control: * information sheet delivered to patients with explanation about the aim of the study,
  * brief interview with the physician about study.

SUMMARY:
Background :

Community-acquired pneumonia (CAP) is a threat in industrialized countries. It represents the 6th cause of death. CAP also frequently associates with other disorders responsible for admission and death. Among bacteria responsible for CAP, Streptococcus pneumonia is a major pathogen that is commonly involved and frequently leads to severe infection and admission. Categories at risk for this pathogen have been determined, and can be proposed anti-pneumococcal vaccination (APV) that efficiently and safely protects from this microorganism.

In the context of US health services, monocenter pilot experiences have reported improvement of pneumococcal prophylaxis implementing vaccination procedure at ED. A study that set in New Mexico (2003) reported a significant increase in APV (from 18% to 84%) when patients at risk were proposed vaccination at ED. To obtain these results, medical students were specifically trained and dedicated to screen and vaccinate against St. pneumoniae. Another single center trial (Tennessee, 2007) for APV at ED obtained an improvement (from 38.8 to 45.4%) when physicians were alerted for pneumococcal risk by the software they usually utilized at bedside. However these experiences remain sparse as additional dedicated resources are required or patients and attending ED physicians can be reluctant to proceed to vaccination at ED.

Mobile phone and derived communication modalities are current vectors to deliver information in several fields including education and medicine. Initially used in developing countries, short-message services (SMS) have improved behaviour of patients in various medical areas. In France, the investigators have observed that most patients above 50 years of age admitted after ED visit are equipped with mobile phone and can receive alerts by SMS.

These observations prompt us to propose a multifaceted procedure to improve APV after ED visit in at-risk patients, combining structured oral interview, written information and SMS as reminders.

Purpose : The investigators hypothesized that

* a multifaceted intervention to promote anti-pneumococcal vaccination combining a structured oral interview, a written information to patient and his/her general practitioner, and a series of 3 SMS,
* improves anti-pneumococcal vaccination at 6 months,
* in at-risk patients (65+ years) visiting the emergency department. In order to answer this question, the investigators designed an interventional prospective multicenter randomized study (cluster).

ELIGIBILITY:
Inclusion Criteria:

* patients 65-year old and above,
* benefit from French or Monaco social security a social security.

Exclusion Criteria:

* refuse to participate,
* no possibility to receive SMS,
* impaired cognitive functions and mental status precluding understanding of the study,
* anticipated barriers precluding adequate follow-up (ex. homeless),
* previous APV,
* contraindication to APV,
* do not understand/read French.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patient aged 65 years or over who is not vaccinated against pneumoccocus virus during consultation with medical emergencies
Sampling Method: Probability Sample
Enrollment: 1475 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Impact of a multifaceted procedure at ED visit on anti-pneumococcal vaccination. (APV) at 6-month. Evaluation criteria : Δ percentage (%) of APV vaccination at 6-month | 6 month

SECONDARY OUTCOMES:
On Flu vaccination at 6-month Δ percentage (%) | 6 month
  number of patients receiving vaccination against flu at 6-month. This issue will be collected by phone (patient, relative or general practioner). This will be a declarative data
On episodes of respiratory tract infections requiring antibiotics or admission at 6-month Δ (absolute number of events) | 6 month
  number of patients who experienced respiratiory tract infection requiring antibiotics or admission. This issue will be collected by phone at 6-month (patient, relative or general practioner). This will be a declarative data
On death at 6- and 12-month (absolute number of events) | 6 month
On death related to infection at 6- and 12-month (absolute number of events) | 6 month
Psychosocial evaluation of patients and acceptance / refusal of vaccination | 6 month
  The patient will fil a Psychosocial evaluation questionnaire during the ED visit. To achieve this issue, we will use the socio-economic indicators mobilized in investigations in social epidemiology: sex, age, education, occupation, housing, income and household size. This composite questionnaire will be used for qualitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yann-Erick CLAESSENS, MD-PHD, Study Director — Centre Hospitalier Princesse Grace; Xavier DUVAL, MD-PHD, Study Director — Groupe Hospitalier Bichat Claude-Bernard; José LABARERE, MD, Study Director — University Hospital, Grenoble; Jocelyn RAUDE, PHD, Study Director — Ecole des Hautes Etudes en Santé Publique
Locations (18):
- France (17):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Paul Ardier, Issoire
  - AP-HM - Hôpital Nord, Marseille
  - AP-HM - La Timone, Marseille
  - HIA Laveran, Marseille
  - Centre Hospitalier La Palmosa, Menton
  - Centre Hospitalier Universitaire de Nice, Nice
  - Centre Hospitalier Louis Giorgi, Orange
  - Hôpital Lariboisière, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Bichat-Claude Bernard, Paris
  - Hôpital Tenon, Paris
  - Hôpital Cochin, Paris
  - Centre hospitalier de Saint-Denis, Saint-Denis
  - Centre Hospitalier de Vaison-la-Romaine, Vaison-la-Romaine
  - Centre Hospitalier Jules Niel, Valréas
  - Centre Hospitalier Jacques Lacarin, Vichy
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No